CLINICAL TRIAL: NCT05990348
Title: Estimation of the Diaphragm Electrical Activity and Intercostal Thickening Fraction During Different Pattern of Mechanical Ventilation: PSV Versus NAVA
Acronym: InterThick
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, SPINAZZOLA GIORGIA, Medical Doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4856
Record Dates: First submitted 2023-02-24; First posted 2023-08-14 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Respiratory Failure; Weaning Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: difficult weaning patients — intercostal thickening fraction values during PSV and NAVA modalities in patients with difficult weaning from MV admitted in ICU.

SUMMARY:
the introduction of new MV modalities has shown promising results in reducing the incidence of weaning failure, mainly due to a more physiologic approach which allows respiratory muscle preservation. Among them, the Neurally Adjust Ventilatory Assist (NAVA) seemed to be associated with lower incidence of weaning failure and subsequent duration of mechanical ventilation, compared to standard modalities like the Pressure Support Ventilation (PSV) . Moreover, NAVA allows the evaluation of the diaphragm electrical activity (EAdi), an index of diaphragmatic neural respiratory drive. However, no study has compared TFic values during PSV and NAVA modalities in patients with difficult weaning from MV admitted in ICU.

DETAILED DESCRIPTION:
Respiratory muscles dysfunction is one of the main causes leading to failure of weaning from mechanical ventilation (MV) in critically ill patients. Muscular activity is important during the inspiratory phase of ventilation, which is mainly due to diaphragm and external intercostal muscles. Diaphragm dysfunction is frequent among critically ill patients and ranges from 33 to 95% . Although several indexes have been investigated to help clinician in identifying its disturbance, their clinical value is controversial . External intercostal muscles dysfunction epidemiology is unknown because of lack of non-invasive tool to investigate such condition. However, the echography assessment of intercostal muscles thickening fraction (TFic) has shown promising results in this field as a non-invasive tool to assess inspiratory muscle function and predict weaning failure .

On the other hand, the introduction of new MV modalities has shown promising results in reducing the incidence of weaning failure, mainly due to a more physiologic approach which allows respiratory muscle preservation. Among them, the Neurally Adjust Ventilatory Assist (NAVA) seemed to be associated with lower incidence of weaning failure and subsequent duration of mechanical ventilation, compared to standard modalities like the Pressure Support Ventilation (PSV) [. Moreover, NAVA allows the evaluation of the diaphragm electrical activity (EAdi), an index of diaphragmatic neural respiratory drive . A recent study suggests that EAdi and derived parameters, may be helpful to predict weaning failure in chronic obstructive pulmonary disease (COPD) patients .

However, no study has compared TFic values during PSV and NAVA modalities in patients with difficult weaning from MV admitted in ICU.

the aim of this study will be the comparison of TFic values during PSV and NAVA modalities in patients with difficult weaning from MV admitted in ICU and the assessment of the inspiratory effort parameters and the occurrence of respiratory asynchrony in patients with difficult weaning from MV admitted in ICU.

ELIGIBILITY:
Inclusion Criteria:

* patients who have failed at least one weaning attempt
* mechanical ventilation for at least 24 hours

Exclusion Criteria:

* Pregnancy
* Obesity (Body Mass Index > 35 kg/m2)
* Contraindication to the insert of a nasogastric tube
* Neuromuscular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients on mechanical ventilation (MV) for at least 24 hours, who have failed at least one weaning attempt, hospitalized at the Intensive Care Unit of Fondazione Policlinico Universitario A. Gemelli IRCCS.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
intercostal thickening fraction | From date of enrollment until the date of extubation (up to seven days)
  intercostal thickening fraction values during PSV and NAVA

CONTACTS AND LOCATIONS:
Locations (1):
- Giorgia Spinazzola, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided
We will assess the availability of data based on the results

REFERENCES:
- [Result] Abdelwahed WM, Abd Elghafar MS, Amr YM, Alsherif SEI, Eltomey MA. Prospective study: Diaphragmatic thickness as a predictor index for weaning from mechanical ventilation. J Crit Care. 2019 Aug;52:10-15. doi: 10.1016/j.jcrc.2019.03.006. Epub 2019 Mar 15. No abstract available. PMID 30904733
- [Result] Spadaro S, Grasso S, Mauri T, Dalla Corte F, Alvisi V, Ragazzi R, Cricca V, Biondi G, Di Mussi R, Marangoni E, Volta CA. Can diaphragmatic ultrasonography performed during the T-tube trial predict weaning failure? The role of diaphragmatic rapid shallow breathing index. Crit Care. 2016 Sep 28;20(1):305. doi: 10.1186/s13054-016-1479-y. PMID 27677861
- [Result] Goligher EC, Dres M, Patel BK, Sahetya SK, Beitler JR, Telias I, Yoshida T, Vaporidi K, Grieco DL, Schepens T, Grasselli G, Spadaro S, Dianti J, Amato M, Bellani G, Demoule A, Fan E, Ferguson ND, Georgopoulos D, Guerin C, Khemani RG, Laghi F, Mercat A, Mojoli F, Ottenheijm CAC, Jaber S, Heunks L, Mancebo J, Mauri T, Pesenti A, Brochard L. Lung- and Diaphragm-Protective Ventilation. Am J Respir Crit Care Med. 2020 Oct 1;202(7):950-961. doi: 10.1164/rccm.202003-0655CP. PMID 32516052
- [Result] Schmidt M, Kindler F, Cecchini J, Poitou T, Morawiec E, Persichini R, Similowski T, Demoule A. Neurally adjusted ventilatory assist and proportional assist ventilation both improve patient-ventilator interaction. Crit Care. 2015 Feb 25;19(1):56. doi: 10.1186/s13054-015-0763-6. PMID 25879592